CLINICAL TRIAL: NCT00432068
Title: A Phase I , Open Label, Single Center, Dose Escalation Study to Assess the Pharmacokinetics, Safety and Tolerability of a Single Dose of a New Extended Long-acting Formulation of Octreotide Pamoate Administered i.m. in Healthy Cholecystectomized Volunteers
Brief Title: Open Label Study of a Single Dose of a New Extended Long Acting Formulation of Octreotide Pamoate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995K2101
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Cholecystectomized
Keywords: Healthy volunteers; octreotide pamoate; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Octreotide pamoate (Experimental)
  Interventions: Drug: Octreotide pamoate

INTERVENTIONS:
Drug: Octreotide pamoate

SUMMARY:
This study will assess the pharmacokinetic profile, safety and tolerability of an octreotide extended long-acting formulation after a single dose in humans. It will investigate the profile of a single dose of drug in a healthy volunteer subject in order to understand the timing and extent of fluctuations in octreotide concentrations in the blood with this formulation, the relationship of drug concentration with dose, and how long the drug remains in the body system.

ELIGIBILITY:
Inclusion criteria:

* Male or female from 18-60 years of age, cholecystectomized at least 4 months prior to the start of the study.
* In a good health as determined by past medical history, physical examination, vital signs, electrocardiogram and laboratory tests at screening
* Body mass index within 19-29 kg/m2
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion criteria:

* Any clinically significant abnormal laboratory values at screening, or evidence of clinically significant abnormal findings at the physical exam at screening, or significant illness within 2 weeks prior to dosing
* A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or untreated)
* History of clinically significant drug allergy, history of atopic allergy, history or clinical evidence of pancreatic injury or pancreatitis, clinical evidence of liver disease or liver injury , history or presence of impaired renal function, or history of urinary obstruction or difficulty urinating
* History of immunocompromise, including a positive HIV
* Known positive hepatitis B or C surface antigen (HBsAg) or Hepatitis C test result (anti-HCV)
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays at screening
* Female subjects who are pregnant or lactating, or are of childbearing potential and without a medically acceptable and highly effective method for birth control.
* Demonstrating intolerance to octreotide at baseline
* Any subject who has a known history of diabetes mellitus in parents or grandparents.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of a single dose of an extended long-acting formulation of octreotide pamoate | 30min, 1, 2, 3, 4, 6, 8, 10, 12 and 24hrs post dose; Thereafter every 5 days for the first 40 days and every 7 days until study completion, 5 to 10 mins apart.
Safety and tolerability assessed by physical exam, ecg, laboratory data and adverse event monitoring | 48 hrs post study drug administration

SECONDARY OUTCOMES:
To determine the relative bioavailability of a single dose of an extended long-acting formulation of octreotide pamoate | 30min, 1, 2, 3, 4, 6, 8, 10, 12 and 24hrs post dose. Thereafter every 5 days for the first 40 days and every 7 days until study completion, 5 to 10 mins apart

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (6):
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Wavre-Gelgique
- France (3):
  - Novartis Investigative Site, Lagord
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
- Novartis Investigative Site, Verona, Italy

IPD SHARING:
Plan to Share IPD: No